CLINICAL TRIAL: NCT06472739
Title: The Effect of GM-CSF to Preventing Oral Mucositis for Patients With Nasopharyngeal Carcinoma Receiving Radiotherapy: A Single-center, Phase II, Randomized Trial
Brief Title: The Effect of GM-CSF to Preventing Oral Mucositis for Patients With Nasopharyngeal Carcinoma Receiving Radiotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GM-CSF for OM
Record Dates: First submitted 2023-08-30; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: GM-CSF
Keywords: Nasopharyngeal Carcinoma; GM-CSF; oral mucositis
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Stomatitis | interventions — Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GM-CSF group (Experimental): Patients use GM-CSF mouthwash four times per day during radiotherpay.
  Interventions: Drug: GM-CSF
- Convertional care group (No Intervention): Patients receive convertional care during radiotherapy.

INTERVENTIONS:
Drug: GM-CSF — GM-CSF mouthwash four times per day at radiotherapy initiate, during the whole radiotherapy phase
  Arms: GM-CSF group

SUMMARY:
To evaluate the efficacy of GM-CSF to preventing oral mucositis for patients with nasopharyngeal carcinoma receiving radiotherapy.

DETAILED DESCRIPTION:
Patients of GM-CSF group receive GM-CSF washmouth four times a day during radiotherapy. Control arm receive conventioanl care during radiotherapy. Visual signs of radiation or chemotherapy-induced mucosal damage were independently assessed during the course of RT by a radiation oncologist or other trained study personnel. The incidence of severe oral mucositis, the severe oral mucositis last time, quality of life between the two arms would be calculated.

ELIGIBILITY:
Inclusion Criteria:

* a. Patients with histologically confirmed non-keratinizing nasopharyngeal carcinoma (including differentiated type and undifferentiated type, world health organization [WHO] II or III).

  b. Original clinical staged as II-IVa (according to the 8 th AJCC edition) c. Male or female who are not pregnant. d. No evidence of distant metastasis (M0). e. Age between 18-65 years. f. WBC≥4×109/L, PLT≥100×109/L, HGB≥90g/L. g. Normal liver function test: Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) <1.5×upper limit of normal (ULN) concomitant with alkaline phosphatase (ALP) ≤2.5×ULN, and bilirubin ≤ULN.

  i. With normal renal function test (creatinine clearance rate≥60 ml/min or creatinine< 1.5×ULN.

  j. The Eastern Cooperative Oncology Group (ECOG) Performance status less or equal to 1.

  k. Patients must be informed of the investigational nature of this study and give written informed consent.

  l. Patients receive induction chemotherapy plus concurrent chemoradiotherpy or concurrent chemoradiotherapy, or radiotherapy alone.

Exclusion Criteria:

* Age <18 or >65years. c. With clinical stage of I or IVb (according to the 8 th AJCC edition). d. Patients with tumor recurrence or distant metastasis. e. Prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer.

  f. History of previous radiotherapy (except for non-melanomatous skin cancers outside intended RT treatment volume).

  g. Prior chemotherapy or surgery (except diagnostic) to primary tumor or nodes.

  h. Pregnancy or lactation (consider pregnancy test in women of child-bearing age and emphasize effective contraception during the treatment period).

  i. Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, acute exacerbation of chronic obstructive pulmonary disease or other respiratory illness requiring admission to hospital, renal disease, chronic hepatitis, diabetes with poor control (fasting plasma glucose >1.5×ULN), and mental disturbance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-08-15 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
The incidence of severe oral mucositis(grade 3+) | During radiotherapy, up to 1.5 months.
  To evaluate the incidence of severe oral mucositis between the two arms.

SECONDARY OUTCOMES:
Acute toxicities | One month.
  The incidence rates of acute toxicities during treatment, evaluted by CTCAE Version5.0.
The last time of ≥3 grade oral mucositis | 1 months after radiotherapy
  The time from first observed ≥3 grade oral mucositis to first observed oral mucositis decrease to less than grade 3
Daily questionaire of oral mucositis (OMDQ) | 1 months after radiotherapy
  Patients are required to finish daily questionaire of oral mucositis by visual signs
Quality of life(QOL) | 1 months after radiotherapy
  QOL is calculated by QLQ-C30.

CONTACTS AND LOCATIONS:
Overall Officials: Qiu Yan Chen, Dr, Study Chair — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No